CLINICAL TRIAL: NCT06471335
Title: Fetal Alcohol Spectrum Disorder (FASD): Clinical Description and Search for Epigenetic Biomarkers for Diagnostic Purposes.
Brief Title: Fetal Alcohol Spectrum Disorder : Clinical Description and Search for Epigenetic Biomarker (EPI-TSAF)
Acronym: EPI-TSAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-A00029-38
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Fetal Alcohol Spectrum Disorders
Keywords: Fetal Alcohol Spectrum Disorders; epigenetic; microRNA
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders

STUDY DESIGN:
Intervention Model Description: This research is descriptive and monocentric research.
  * retrospective on the clinical description of the 182 Fetal Alcohol Spectrum Disorder patients
  * prospective on the microRNAs part with 18 patients in Fetal Alcohol Spectrum Disorder group and 18 people in the control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients Fetal Alcohol Spectrum Disorder (Experimental): Patients with Fetal Alcohol Spectrum Disorder, male an female, aged 0 to 18 inclusive.
  Interventions: Diagnostic Test: Extraction of microRNAs extracted from plasma (4 ml recovered as part of treatment); Diagnostic Test: Extraction of microRNAs extracted from bucal swabs (act added for research).
- Participants without Fetal Alcohol Spectrum Disorder (Active Comparator): Participants without Fetal Alcohol Spectrum Disorder, male an female, aged 0 to 18 inclusive.
  Interventions: Diagnostic Test: Extraction of microRNAs extracted from bucal swabs (act added for research).

INTERVENTIONS:
Diagnostic Test: Extraction of microRNAs extracted from plasma (4 ml recovered as part of treatment) — Comparison of these micro RNAs with the micro RNAs extracted from oral swabs (in Fetal Alcohol Spectrum Disorder group)
  Arms: Patients Fetal Alcohol Spectrum Disorder
Diagnostic Test: Extraction of microRNAs extracted from bucal swabs (act added for research). — Comparison of the microRNAs extracted from the oral swabs of the Fetal Alcohol Spectrum Disorder group with the microRNAs extracted from the oral swabs of the without Fetal Alcohol Spectrum Disorder group

SUMMARY:
The goal of this clinical trial is to carry out a clinical description of a Reunionese series of patients (aged 0 to 18 inclusive) with Fetal Alcohol Spectrum Disorders followed up in the Genetics Department of the University Hospital in Reunion Island The aim is also to identify a specific "epigenetic signature" for Fetal Alcohol Spectrum Disorder, in order to provide early diagnostic markers, determine the origin of the microRNAs identified and study the phenotypic-epigenetic relationship (microRNAs).

This research is descriptive and monocentric.

* retrospective on the clinical description of 182 Fetal Alcohol Spectrum Disorderpatients
* prospective on the microRNAs part, with 18 patients in the Fetal Alcohol Spectrum Disorder group and 18 in the control group (participants without Fetal Alcohol Spectrum Disorder).

For the 18 patients in the Fetal Alcohol Spectrum Disorder group, the doctor will take a blood sample (for genetic testing) during a scheduled consultation. A remaining 4 ml of blood will be collected for research purposes (Fetal Alcohol Spectrum Disorder group only). A buccal smear will also be taken for research.

For the 18 participants in the control group (healthy participants of the same age and sex as the Fetal Alcohol Spectrum Disorder group), only a buccal smear will be taken for research purposes during a consultation.

ELIGIBILITY:
Inclusion Criteria:

Fetal Alcohol Spectrum Disorder group :

* born in Reunion
* aged between 0 and 18 years old
* Having been exposed to alcohol during the prenatal period
* Have a diagnosis of Fetal Alcohol Spectrum Disorder by a referring physician

Control group :

* born in Réunion
* aged between 0 and 18 years old
* Be matched on the age and sex of the Fetal Alcohol Spectrum Disorder children sampled (n=18)
* Not having been exposed to alcohol during the prenatal period
* Not having been diagnosed with FASD
* Not have congenital malformations
* Not have neurodevelopmental disorders

Exclusion Criteria:

Fetal Alcohol Spectrum Disorder group :

* patients with Fetal Alcohol Spectrum Disorder who also present another genetic syndrome.

Control group :

- people who are not matched on the age and sex of the Fetal Alcohol Spectrum Disorder patients sampled

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 188 (Actual)
Dates: Start 2024-06-12 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-23 (Actual)

PRIMARY OUTCOMES:
Clinical description of a series of Fetal Alcohol Spectrum Disorder patients from Reunion Island (part 1) | 6 months
  Description of :
  * maternal alcohol consumption in the prenatal period and paternal alcohol consumption in the preconception period :
  * duration (in month)
  * type (Beer, wine, strong alcohol, Multiple)
  * frequency (DAILY/ WEEK/ WEEKEND/ FESTIVAL-OCCASIONAL/ SINGLE EPISODE )
  * stage of exposure (Trimester : 1/2/ ≤ 2 /3/≤ 3)
  * other associated toxicants : tobacco, cannabis, medications (Yes/ no/ suspicion)
  * the course of the pregnancy and childbirth :
  * age of the mother (in years)
  * term of delivery (FULL-TERM/ MEDIUM PREMATURITY/ HIGH PREMATURITY/ VERY HIGH PREMATURITY)
  * trimester of discovery of the pregnancy (trimester : 1, 2, 3)
  * socio-family data
  * family situation (ADOPTION/ MOTHER/ PARENTS/ FATHER)
  * type of placement (FOSTER FAMILY/ HOME/ ADOPTIVE FAMILY/ THIRD PARTY/ NURSERY)
  * age of placement (in years)
Clinical description of a series of Fetal Alcohol Spectrum Disorder patients from Reunion Island (part2) | 6 months
  Description of :
  * data from the medical and genetic assessment
  * congenital malformations (Yes/ No)
  * hearing assessment (Normal/ abnormal),
  * Chromosome analysis on a DNA chip (Normal/ abnormal),
  * fragile X (Normal/ abnormal)
  * data from the neuropsychological and psychomotor assessment
  * psychomotor delay (Yes/ No)
  * motor impairments (Yes/ No)
  * intellectual disability (Yes/ No) (IQ Value)
  * cognitive impairments (VERY WEAK/ LIMITED/ MEDIUM WEAK/ MEDIUM/ MEDIUM STRONG/ SUPERIOR/ VERY SUPERIOR)
  * oral language, executive functions, behavioral abnormalities (alter/preserve),
  * data from paraclinical examinations :
  * kidney ultrasound, cardiac ultrasound, Magnetic Resonance Imaging (Nomal/ Abnormal)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de la Réunion, Saint-Denis, France

IPD SHARING:
Plan to Share IPD: No